CLINICAL TRIAL: NCT04927052
Title: A Multicenter, Double-Blind, Randomized, Split-Face Study to Evaluate the Safety and Efficacy of Revanesse Shape + With Lidocaine Versus Juvederm Voluma With Lidocaine for the Correction of Age-Related Midface Volume Deficit / Lipoatrophy at 6 and 12 Months Post-treatment
Brief Title: A Study to Evaluate the Safety and Efficacy of Revanesse Shape + With Lidocaine Versus Juvederm Voluma With Lidocaine for the Correction of Age-Related Midface Volume Deficit / Lipoatrophy at 6 and 12 Months Post-treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prollenium Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO 2019-04 CAN
Record Dates: First submitted 2021-06-02; First posted 2021-06-15 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Volume Deficit in the Mid-face

STUDY DESIGN:
Intervention Model Description: A split-face study in subjects seeking to correct mid-face volume deficit. Subjects will be treated with Revanesse Shape + with Lidocaine on one side of the face and Juvederm Voluma with Lidocaine on the other side of the face. The side of the face for each device will be randomly assigned.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Additionally, the Sponsor's staff conducting the study, and members of the administrative team will not have access to individual subjects' treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Revanesse Shape + with Lidocaine (Active Comparator): Revanesse Shape + with Lidocaine is a clear, colorless gel in 1.2 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid and lidocaine 0.3% w/w. Participants had 1 cheek treated with Revanesse Shape + with Lidocaine
  Interventions: Device: Revanesse Shape + with Lidocaine; Device: Juvederm Voluma with Lidocaine.
- Juvederm Voluma with Lidocaine (Active Comparator): Juvederm Voluma with Lidocaine is a clear, colorless gel in 1.0 mL pre-filled syringes formulated to a concentration of 20 mg/mL of stabilized hyaluronic acid and lidocaine 0.3% w/w. Participants had 1 cheek treated with Juvederm Voluma with Lidocaine.
  Interventions: Device: Revanesse Shape + with Lidocaine; Device: Juvederm Voluma with Lidocaine.

INTERVENTIONS:
Device: Revanesse Shape + with Lidocaine — Revanesse Shape + with Lidocaine. Participants had 1 cheek treated with Revanesse Shape + with Lidocaine
Device: Juvederm Voluma with Lidocaine. — Juvederm Voluma with Lidocaine. Participants had 1 cheek treated with Juvederm Voluma with Lidocaine

SUMMARY:
To compare the safety and efficacy profiles of Revanesse Shape + with Lidocaine versus Juvederm Voluma with Lidocaine for subcutaneous and/or supraperiosteal injection to improve appearance through the correction of age-related mid-face volume deficit in patients 22 years of age through 65 years of age.

Midface volume deficit / lipoatrophy (loss of subcutaneous adipose tissue that is most apparent in the face) may be associated with acquired conditions, the aging process, or based on genetic causes.

DETAILED DESCRIPTION:
This is a randomized, multicenter, double blind, split-face study in subjects seeking to correct mid-face volume deficit. Subjects will be treated with Revanesse Shape + with Lidocaine on one side of the face and Juvederm Voluma with Lidocaine on the other side of the face. The side of the face for each device will be randomly assigned. The Evaluating Investigator performing the evaluations and the subject will be blinded to the treatment; injections of the study device will be performed by an unblinded Treating Investigator.

At each visit, the blinded Evaluating Investigator evaluations and subject evaluations of the treated areas will be performed and recorded.

The initial treatment will be done at Visit 1 and a touch-up if necessary at Visit 3/Month 1. One optimal correction touch-up can be administered for subjects who experience asymmetrical cheeks after Visit 5/Month 3 and before Visit 7/Month 12 . The Blinded Evaluating Investigator will confirm the asymmetry with at least a 1-grade difference between cheeks. The touch up will be offered on the under-corrected side with the same product that was initially implanted. In addition, subjects will have a safety follow-up telephone call 3 days (± 2 days) after any optimal correction touch-up to correct asymmetry administered between Visit 5/Month 3 and Visit 7/Month 12.

Subjects will be retreated at the Month 12 Visit if a ≥ 1 grade change or return to baseline of the MMVS scores on one or both sides of the face.

Treatment Phase

* Visit 1 - (Day 1) - Baseline and treatment
* Day 3 (+2/-1 days) - Safety follow-up telephone call
* Visit 2 - Week 2 (Day 14 ± 2 days) - Safety follow-up visit
* Visit 3 - Month 1 (Day 30 ± 2 days) - interim visit, optimal correction touch-up if needed
* If touch up administered at Visit 3:
* Safety follow-up telephone call 3 days after touch-up (± 2 days)
* Visit 3a - Day 14 ± 2 days after touch-up - Safety follow-up visit Safety and Effectiveness Phase
* Visit 4 - Month 2 (Day 60 ± 2 days) - interim visit
* Visit 5 - Month 3 (Day 90 ± 2 days) - interim visit
* Visit 6 - Month 6 (Day 180 ± 4 days) - interim visit Extended Follow-up Phase
* Visit 7 - Month 12 (Day 360 ± 4 days) - interim visit Retreatment if needed
* If Retreatment administered at Visit 7:
* Safety follow-up telephone call 3 days after retreatment (± 2 days)
* Visit 7a - Day 14 ± 2 days after retreatment - Safety follow-up visit
* Visit 8 - Month 15 (Day 450 ± 4 days) - End of Study Visit Optimal Correction Touch-up to correct asymmetry
* Visit 6a - After Visit 5/Month 3 and before Visit 7/Month 12) - optimal correction touch-up to correct asymmetry
* 3 days after touch-up (± 2 days) - Safety follow-up telephone call

Evaluations include:

Medicis Mid-face Volume Scale (MMVS) score Global Aesthetic Improvement Score (GAIS) by subject and Evaluating Investigator Nasolabial Folds Wrinkle Severity Rating Score (WSRS) Safety will be assessed by monitoring adverse events (AEs) at all study visits. In addition, other mid-face safety evaluations including firmness, function (movement), mass formation and sensation will be performed at baseline and follow up visits.

Other evaluations include subject overall satisfaction of facial appearance, subject satisfaction with mid-facial region, subject look of mid-face, subject feel of mid-face, subject self-perception of age, subject happiness with contour/shape of mid-face, subject self confidence, subject recommendation to a friend, and subject self perception of age since baseline.

Other analysis includes subject comfort and Unblinded Treating Investigator Ease of Use assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant, non-breastfeeding women 22 years of age through 65 years of age.
2. Subjects seeking augmentation therapy for the mid-face with a MMVS score of 3 (moderate loss of fullness with slight hollowing) or 4 (substantial loss of fullness in the mid-face area, clearly apparent hollowing) on each side of the face as independently assessed by the blinded Evaluating Investigator and the unblinded Treating Investigator
3. If female and of childbearing potential, a negative urine pregnancy test at Baseline (Day 1) and the subject agrees to use adequate contraception during the study period.
4. Ability to understand and comply with the requirements of the study.
5. Willingness and ability to provide written informed consent.
6. Willing to abstain from any other facial procedures or treatments affecting facial volume deficit at any time during the study

Exclusion Criteria:

1. MMVS score of 1 (fairly full) or 2 (mild loss of fullness) on either side of the face.
2. Women who are pregnant or lactating or anticipate becoming pregnant during the study period.
3. Have ever undergone facial plastic surgery (with the exception of rhinoplasty more than 2 years prior to enrollment), tissue grafting, or tissue augmentation with silicone, fat, or other permanent (Ex: polymethylmethacrylate (Bellafill)), or semi-permanent dermal fillers (Ex: calcium hydroxylapatite (Radiesse®)) or planning to undergo any of these procedures at any time during the study.
4. Have undergone temporary facial dermal filler injections with hyaluronic acid-based fillers within 12 months, porcine-based collagen fillers within 12 months, or neuromodulator injections, mesotherapy, or resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, microneedling or other ablative or non-ablative procedures) within 6 months on the face or neck prior to study entry or planning to undergo any of these procedures at any time during the study.
5. History of use of threads below the lower orbital rim within the preceding 6 months or planning their use at any time during the study
6. History of use of injectable deoxycholate (Kybella®) anywhere on the face or neck within preceding 6 months or planning to undergo treatment at any time during the study
7. Evidence of scar-related disease or delayed healing activity to the mid-face within the past 1 year.
8. Has acute or chronic skin disease or scars at the intended treatment sites.
9. History of keloid formation or hypertrophic scars.
10. History or the presence of any disease that may result in changes in facial contour or edema of the face during the course of the study, (e.g., inflammation, infection, facial psoriasis, herpes zoster, acanthosis, cancer, pre-cancer, actinic keratosis, etc.)
11. Presence of active inflammatory process (skin eruptions such as cysts, pimples, rashes, or hives) or infection on the face.
12. Have severe malocclusion or dentofacial or maxillofacial deformities as judged by the Treating Investigator. Subjects planning to undergo extensive dental procedures such as dental implants, multiple tooth extractions, or oral surgery should not participate. Minor dental procedures such as teeth cleaning and repair of caries are not exclusionary.
13. Is on an ongoing regimen of anticoagulation therapy (e.g., warfarin), thrombolytics, or inhibitors of platelet aggregation
14. Nonsteroidal anti inflammatory drugs (NSAIDs, e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or gingko) within 10 days of undergoing study device injections. Subjects who will withhold such therapy for 10 days before AND after any injection session may participate.
15. Prescription, oral or topical anti-wrinkle products in the treatment area within 90 days prior to treatment and throughout the study. (Use of sunscreens and continued therapy with OTC topical treatments (e.g., alpha hydroxyl acids, glycolic acids, retinoids) are allowed if regimen was established ≥ 90 days prior to treatment).
16. History of allergy, anaphylaxis or hypersensitivity to injectable hyaluronic acid products, local anesthetics of the amide type such as lidocaine, or gram positive bacterial proteins or is planning to undergo desensitization therapy during the study.
17. History or presence of multiple severe allergies or severe allergies manifested by a history of anaphylaxis.
18. History of known streptococcal disease.
19. Immunocompromised, immunosuppressed or current use of immunosuppressive therapy that in the opinion of the investigator precludes participating in the trial.
20. Clinically significant organic disease including cardiovascular, hepatic, pulmonary, neurologic, or renal disease or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator, precludes participation in the trial.
21. History or presence of porphyria
22. Have untreated epilepsy
23. History of connective tissue diseases such as rheumatoid arthritis, systemic lupus erythematosus, polymyositis (PM), dermatomyositis (DM) or scleroderma
24. Have bleeding disorders
25. Presence of wound on the face
26. Received any investigational product within 30 days of signing the ICF.
27. Facial tattoo that may interfere with MMVS evaluation.
28. Presence of facial hair that could interfere with MMVS evaluation. Subjects with facial hair must agree to maintain the same style and length of facial hair throughout the duration of the study.
29. Systemic (oral/injectable) corticosteroids, anabolic steroids or immunosuppressive medications within 30 days prior to treatment and topical steroids on the face within 14 days prior to treatment start and throughout the study.
30. Previous treatment for MVD within the past year.
31. History of malignancy within 5 years of study entry. Subjects with a history of malignancy that has been fully treated without evidence of recurrence for at least five years prior to study entry may participate. (Subjects with a history of basal cell carcinoma or squamous cell carcinoma outside of the treatment area that has been fully removed by surgical means may participate at any time).
32. Currently has a cancerous or pre-cancerous lesion on the treatment area or has had radiation exposure in the treatment area in the last 24 months.
33. The presence of any condition, which in the opinion of the investigator, that makes the subject unable to complete the study per protocol (e.g., subjects not likely to avoid other facial cosmetic treatments, subjects not likely to stay in the study because of other commitments, concomitant conditions or past history; subjects anticipated to be unreliable; or subjects who have a concomitant condition that might confuse or confound study treatments or assessments).
34. The intention to lose a significant amount of weight (more than 10 pounds) during the study.
35. Presence of moderate or severe abnormal rating for firmness or detection of any abnormal mid-face structure, such as a scar or lump at baseline.
36. Presence of abnormal rating in mid-face function with inability to effectively puff cheeks, smile broadly, or chew at baseline.
37. Presence of abnormal rating in mid-face sensation with inability to feel 0.4G monofilament or cotton wisp at any site on the mid-face at baseline
38. Presence of abnormal vision assessments at baseline, e.g., Snellen Acuity Test worse than 20/40 (with corrections, if applicable), abnormal confrontational visual field test, or abnormal ocular motility test).

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Visit 6/Month 6 in the Medicis Mid-face Volume Scale (MMVS) score | Baseline visit to Visit 6/Month 6.
  The blinded evaluating investigator assessed the participant's overall mid-face volume deficit for each cheek using a 4-point photonumeric scale, where: 1=None (fairly full midface) [best] to 4=Substantial (substantial loss of fullness in the mid-face area) [worst]. A negative change from Baseline indicates improvement

SECONDARY OUTCOMES:
Change from baseline to Visit 7/Month 12 in the Medicis Mid-face Volume Scale (MMVS) score | Baseline visit to Visit 7/Month 12
  The blinded evaluating investigator assessed the participant's overall mid-face volume deficit for each cheek using a 4-point photonumeric scale, where: 1=None (fairly full midface) [best] to 4=Substantial (substantial loss of fullness in the mid-face area) [worst]. A negative change from Baseline indicates improvement
Change in the Nasolabial Folds Wrinkle Severity Rating Scale score at Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15 | Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15
  The blinded evaluating investigator assessed the participant's nasolabial folds for each cheek using a 5-point scale, where: 1=Absent (No visible folds) [best] to 5=Extreme (Extremely deep and long folds) [worst]. A negative change from Baseline indicates improvement
Percent of subjects with clinical success at Visit 6/Month 6 where success is defined as a subject with at least a 1-grade improvement from baseline on the Investigator Global Aesthetic Improvement Score (iGAIS). | Baseline visit to Visit 6/Month 6
  Clinical success at Visit 6/Month 6 where success is defined as a subject with at least a 1-grade improvement from baseline on the Investigator Global Aesthetic Improvement Score (iGAIS) a 5-point scale where 1=Worse (the appearance is worse than the original condition) [worst] to 5=Very much improved (optimal cosmetic results) [best].
Percent of subjects with treatment success at Visit 6/Month 6 where success is defined as a subject with at least a 1-grade improvement from baseline on the Patient Global Aesthetic Improvement Score (pGAIS) | Baseline to Visit 6/Month 6
  Clinical success at Visit 6/Month 6 where success is defined as a subject with at least a 1-grade improvement from baseline on the Patient Global Aesthetic Improvement Score (pGAIS) a 5-point scale where 1=Worse (the appearance is worse than the original condition) [worst] to 5=Very much improved (optimal cosmetic results) [best].
Percent of subjects with treatment success at Visit 7/Month 12 where success is defined as a subject with at least a 1-grade improvement from baseline on the Patient Global Aesthetic Improvement Score (pGAIS) | Baseline to Visit 7/Month 12
  Clinical success at Visit 7/Month 12 where success is defined as a subject with at least a 1-grade improvement from baseline on the Patient Global Aesthetic Improvement Score (pGAIS) a 5-point scale where 1=Worse (the appearance is worse than the original condition) [worst] to 5=Very much improved (optimal cosmetic results) [best].

OTHER OUTCOMES:
Subject overall satisfaction of facial appearance for each side of the face | Baseline to Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15and every study visit
  Overall Satisfaction with Facial Appearance will be assessed at all visits and prior to any treatment by the subject using a 100 mm VAS scale from 0 = very unsatisfied (worst) to 100 = very satisfied (best)
Subject satisfaction with mid-facial region for each side of the face | Baseline to Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15
  Subject satisfaction with mid-facial region will be assessed at all visits and prior to any treatment by the subject using a 100 mm VAS scale from 0 = very unsatisfied (worst) to 100 = very satisfied (best)
Subject look of mid-face for each side of the face | Baseline to Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15
  Subject look of mid-face will be assessed at all visits and prior to any treatment by the subject using a 100 mm VAS scale from 0 = very unsatisfied (worst) to 100 = very satisfied (best)
Subject feel of mid-face for each side of the face | Baseline to Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15
  Subject feel of mid-face will be assessed at all visits and prior to any treatment by the subject using a 100 mm VAS scale from 0 = very unsatisfied (worst) to 100 = very satisfied (best)
Self-perception of age for each side of the face | Baseline to Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15
  Self-perception of age will be assessed at all visits and prior to any treatment by the subject using a 100 mm VAS scale from 0 = very unsatisfied (worst) to 100 = very satisfied (best)
Subject happiness with contour/shape of mid-face for each side of the face | Baseline to Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15
  Subject happiness with contour/shape of mid-face will be assessed at all visits and prior to any treatment by the subject using a 100 mm VAS scale from 0 = very unsatisfied (worst) to 100 = very satisfied (best)
Subject self confidence for each side of the face | Baseline to Visit 2/Week 2, Visit 3/Month 1, Visit 4/Month 2, Visit 5/Month 3, Visit 6/Month 6, Visit 7/Month 12 and Visit 8/Month 15
  Subject's self confidence will be assessed at all visits and prior to any treatment by the subject using a 100 mm VAS scale from 0 = very unsatisfied (worst) to 100 = very satisfied (best)
Subject recommendation to a friend for each side of the face | Visit 8/Month 15 or study completion if earlier than Month 15
  Subjects will be asked if they would recommend the treatment to a friend
Subject self perception of age since baseline for each side of the face | Visit 8/Month 15 or study completion if earlier than Month 15
  Subjects will be asked their self perception of age since baseline on a 4 point scale with 1 = Not younger than my actual age (worst) to 4=More than 10 years younger than my actual age (best)

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Laser Rejuvenation, Calgary, Alberta
  - Alpha Research/Lucere Dermatology, Edmonton, Alberta
  - Dermetics, Burlington, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - Bertucci MedSpa, Woodbridge, Ontario
  - Victoria Park Medispa Laval, Laval, Quebec
  - Erevna Innovations, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: No